CLINICAL TRIAL: NCT00799487
Title: Double-Blind, Randomized, Placebo-Controlled, Crossover Study Evaluating the Academic, Behavioral and Cognitive Effects of CONCERTA on Older Children With ADHD (The ABC Study)
Brief Title: CONCERTA Lab School Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR015118; NCT00799487; 2015-001042-28 (EudraCT Number)
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- 1 (Experimental): CONCERTA (methylphenidate HCl) or placebo Optimal Subject Dose (18mg-54mg) once daily during Lab School Day #1 with placebo on Day #2
  Interventions: Drug: CONCERTA (methylphenidate HCl) or placebo
- 2 (Experimental): CONCERTA (methylphenidate HCl) or placebo Optimal Subject Dose (18mg-54mg) once daily during Lab School Day #2 with placebo on Day #1
  Interventions: Drug: CONCERTA (methylphenidate HCl) or placebo

INTERVENTIONS:
Drug: CONCERTA (methylphenidate HCl) or placebo — Optimal Subject Dose (18mg-54mg) once daily during Lab School Day #1 with placebo on Day #2
  Arms: 1
Drug: CONCERTA (methylphenidate HCl) or placebo — Optimal Subject Dose (18mg-54mg) once daily during Lab School Day #2 with placebo on Day #1
  Arms: 2

SUMMARY:
The purpose of this trial is to determine if the study medication, CONCERTA (methylphenidate HCl), is safe and effective in improving academic performance and behavior in children with Attention Deficit Hyperactivity Disorder (ADHD) when compared to placebo.

DETAILED DESCRIPTION:
The hypothesis is that CONCERTA (methylphenidate HCl) is safe and effective in improving academic performance and behavior in children with ADHD when compared to placebo as demonstrated using specified study measures. This is a double-blind (neither participant nor investigator knows the name of the assigned study drug), randomized (study drug assigned by chance), placebo-controlled, crossover study evaluating the academic, behavioral and cognitive effects of CONCERTA (methylphenidate HCl) on older children with ADHD This means that all eligible children will receive treatment with methylphenidate HCl throughout the study (the titration and assessment periods) and inactive pill (placebo) on 1 of the 2 laboratory classroom days. On the other laboratory classroom day they will receive their regular dose of CONCERTA (methylphenidate HCl). The primary efficacy variable in this study is the Permanent Product Math Test (PERMP) attempted score. Secondary Measures include: SKAMP (Swanson, Kotkin, Agler, M-Flynn, and Pelham), tests of inattention, reading fluency and comprehension, and memory. Assessments will be completed during each of the laboratory assessment days (12.5 hours). Participants will be assessed for adverse events throughout the study. Patients will initiate treatment with oral CONCERTA (methylphenidate HCl) 18 mg at baseline and continue morning dosing with increases every 3 to 7 days until an optimal dose is achieved, up to the maximum of 54 mg/day. Eligible patients will remain in the study for a maximum of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosis of all subtypes (except Not Otherwise Specified)
* Patients with total or subscale Attention Deficit Hyperactivity Disorder Rating Scale (ADHD RS-IV) scores > =90th percentile relative to the general population of children by age and gender
* Patients currently receiving ADHD medication must be inadequately managed on their current stimulant dose and meet this criteria at the screening visit
* Ability to read and understand English
* Ability to attend school regularly

Exclusion Criteria:

* Estimated Full Scale IQ score of 80 or below, Severe Learning Disability
* History of or current, primary diagnosis of: severe anxiety disorder, conduct disorder, psychotic disorders, Pervasive Developmental Disorder, Eating Disorder, Obsessive-Compulsive Disorder, Sleep Disorder, Major Depressive Disorder, Bipolar Disorder, Substance Use Disorder, Chronic Tic Disorder, personal or family history of Tourette's Syndrome
* Weight < 3rd percentile for age
* History of hospitalization for treatment of a mood, anxiety, or psychotic disorder
* History of failed response to methylphenidate

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2009-01-02 (Actual); Primary Completion 2009-06-26 (Actual); Study Completion 2009-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC
Locations (3):
- United States (3):
  - Little Rock, Arkansas
  - Las Vegas, Nevada
  - Durham, North Carolina

REFERENCES:
- See also: Double-Blind, Randomized, Placebo-Controlled, Crossover Study Evaluating the Academic, Behavioral and Cognitive Effects of CONCERTA on Older Children with ADHD — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=83&filename=CR015118_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Randomized: Children who started dose adjustment period, but were not randomized
- Placebo/Concerta: Children randomized to receive Placebo at lab school day 1 and an individualized, optimal dose of Concerta (18mg, 36mg, or 54mg tablet) once daily at lab school day 2
- Concerta/Placebo: Children randomized to receive an individualized, optimal dose of Concerta (18mg, 36mg, or 54mg tablet) once daily at lab school day 1 and Placebo at lab school day 2
Period: Dose Adjustment Period
Arm/Group | Not Randomized | Placebo/Concerta | Concerta/Placebo
Started | 21 | 34 | 34
Completed | 0 | 34 | 34
Not Completed | 21 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Optimal Dose Not Achieved | 8 | 0 | 0
Not completed — Investigator Discretion | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Parent to home school child (exclusion) | 1 | 0 | 0
Not completed — Child too young (exclusion) | 1 | 0 | 0
Not completed — Missed laboratory day 1 | 1 | 0 | 0
Not completed — ADHD RS-IV rating scale >85th percentile | 2 | 0 | 0
Period: Double-Blind Assessment Period
Arm/Group | Not Randomized | Placebo/Concerta | Concerta/Placebo
Started | 0 | 34 | 34
Completed | 0 | 33 | 32
Not Completed | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Subject was out of the state | 0 | 0 | 1
Not completed — Overslept and missed lab day 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Concerta: Children randomized to receive Placebo at lab school day 1 and Concerta lab school day 2
- Concerta/Placebo: Children randomized to receive Concerta at lab school day 1 and Placebo at lab school day 2
- Total: Total of all reporting groups
Arm/Group | Not Randomized | Placebo/Concerta | Concerta/Placebo | Total
Number analyzed (Participants) | 21 | 34 | 34 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.0 (1.00) | 10.1 (1.07) | 10.4 (0.99) | 10.2 (1.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 | 9 | 29
  Male | 15 | 20 | 25 | 60
Region of Enrollment [Number; unit: participants]
  USA | 21 | 34 | 34 | 89

OUTCOME MEASURES:

1. Primary Outcome: Hour 4 Permanent Product Math Test Attempted Score (PERMP-Attempted)
Description: PERMP (range: 0, 400) is a measure of academic productivity. These seatwork math tasks provide an objective measure of attention and accuracy in calculations. The level of difficulty is established on a screening math pretest. The subsequent laboratory school day assessments employed a series of 10-minute math tests (5 pages of 80 math problem each for a total of 400 problems available). Children were graded on the number of attempted problems. A higher number of problems attempted was indicative of greater attention to detail (higher score is preferable.)
Time Frame: Hour 4 of the Double-Blind Assessment Period Lab School Day
Population: No randomized children were included at this time point. The number of children treated with placebo is based on 68 children minus 3 children who did not crossover and minus 1 child who dropped out before laboratory day 2. The number of children treated with CONCERTA is based on 68 children minus 1 child who dropped out before laboratory day 2.
Measure: Mean (Standard Deviation); unit: Problems attempted
Groups:
- Placebo: Children randomized to receive Placebo at lab school day 1 or lab school day 2
- Concerta: Children randomized to receive Concerta at lab school day 1 or lab school day 2
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Problems attempted |  | 88.0 (39.79) | 116.1 (38.99)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-values were determined by using a repeated measures mixed model with actual value as the dependent variable with terms for treatment, time, treatment by time interaction, period, sequence, and baseline score; LS Mean Difference = -27.3, 95% CI 2-sided [-34.4 to -20.2] — Placebo minus Concerta

2. Primary Outcome: Hour 4 Permanent Product Math Test Correct Score (PERMP-Correct)
Description: PERMP (range: 0, 400) is a measure of academic productivity. These seatwork math tasks provide an objective measure of attention and accuracy in calculations. The level of difficulty is established on a screening math pretest. The subsequent laboratory school day assessments employed a series of 10-minute math tests (5 pages of 80 math problem each for a total of 400 problems available). Children were graded on the number of correct problems. A higher number of problems correct, of those attempted, was indicative of greater accuracy.
Time Frame: Hour 4 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Problems correct
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Problems correct |  | 84.0 (39.93) | 112.8 (39.60)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -28.0, 95% CI 2-sided [-35.1 to -20.8] — Placebo minus Concerta

3. Secondary Outcome: Hour 4 Swanson, Kotkin, Alger, M-Flynn and Pelham Scale for Deportment (SKAMP-Deportment)
Description: The SKAMP scale measures the manifestations of ADHD using an independent observer (teacher) rating of children impairment in classroom behavior. The SKAMP-Deportment (SKAMP-D) (range: 0,36) is a sum of ratings on 6 deportment items (interacting with other children, interacting with adults, remaining quiet, staying seated, complying with the teacher's directions, and following the classroom rules). Each item was rated on a 7-point impairment scale (0=normal, 6=maximum impairment), with higher scores indicating more severe symptoms.
Time Frame: Hour 4 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 8.0 (6.54) | 3.1 (3.65)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 5.0, 95% CI 2-sided [3.4 to 6.6] — Placebo minus Concerta

4. Secondary Outcome: Hour 4 Swanson, Kotkin, Alger, M-Flynn and Pelham Scale for Attention (SKAMP-Attention)
Description: The SKAMP scale measures the manifestations of ADHD using an independent observer (teacher) rating of children impairment in classroom behavior. The SKAMP-Attention (SKAMP-A) (range: 0, 42) is a sum of the ratings on 7 attention items (getting started, sticking with tasks, attending to an activity, making activity transitions, completing assigned tasks, performing work accurately, and being neat and careful while writing or drawing). Each item was rated on a 7-point impairment scale (0=normal, 6=maximum impairment), with higher scores indicating more severe symptoms.
Time Frame: Hour 4 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 10.1 (5.51) | 5.6 (3.69)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 4.5, 95% CI 2-sided [3.2 to 5.8] — Placebo minus Concerta

5. Secondary Outcome: Hour 4 Swanson, Kotkin, Alger, M-Flynn and Pelham Scale for Composite (SKAMP-Composite)
Description: The SKAMP scale measures the manifestations of ADHD using an independent observer (teacher) rating of child impairment in classroom behavior. A composite score (range: 0, 78) for the SKAMP variable (13 items total) was obtained by summing the SKAMP-D and SKAMP-A subscale scores. A lower score was preferable, as a higher score represented greater behavioral impairment.
Time Frame: Hour 4 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo: Chidren randomized to receive Placebo at lab school day 1 or lab school day 2
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 18.1 (10.61) | 8.7 (6.10)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 9.5, 95% CI 2-sided [6.9 to 12.0] — Placebo minus Concerta

6. Secondary Outcome: Hour 5.5 Test of Variables of Attention (TOVA) ADHD Score
Description: The TOVA is a computerized, visual continuous performance test which provides measures of attention. The stimulus, presented for 100 milliseconds (ms) at the rate of 30 per minute, is a computer-presented square containing a square hole near the top (target) or bottom (non-target) edge. The first half of the TOVA requires that the child sustain attention while the second half requires inhibition of response to a non-target (observed range: -15.2, 5.2). An ADHD score of less than -1.80 is suggestive of ADHD.
Time Frame: Hour 5.5 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | -4.19 (3.563) | -0.68 (3.672)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -3.51, 95% CI 2-sided [-4.27 to -2.74] — Placebo minus Concerta

7. Secondary Outcome: Hour 5.5 Test of Variables of Attention (TOVA) Reaction Time (Msec)
Description: The TOVA is a computerized, visual continuous performance test which provides measures of attention. The stimulus, presented for 100 milliseconds (ms) at the rate of 30 per minute, is a computer-presented square containing a square hole near the top (target) or bottom (non-target) edge. The first half of the TOVA requires that the child sustain attention while the second half requires inhibition of response to a non-target. Mean response latency in msecs (observed range: -75.4, 129.5). Higher score indicates faster reaction time.
Time Frame: Hour 5.5 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliseconds (msecs)
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Milliseconds (msecs) |  | 75.23 (26.740) | 93.21 (32.619)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -17.58, 95% CI 2-sided [-23.72 to -11.45] — Placebo minus Concerta

8. Secondary Outcome: Hour 5.5 Test of Variables of Attention(TOVA) Reaction Time Variability (Standard Deviation in Milliseconds (Msecs))
Description: The TOVA is a computerized, visual continuous performance test which provides measures of attention. The stimulus, presented for 100 milliseconds (ms) at the rate of 30 per minute, is a computer-presented square containing a square hole near the top (target) or bottom (non-target) edge. The first half of the TOVA requires that the child sustain attention while the second half requires inhibition of response to a non-target. SD of response times (msecs) (observed range: -177.6, 132.9). Higher score indicates less variability.
Time Frame: Hour 5.5 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Placebo: Children randomized to receive Placebo at lab school day 1 or at lab school day 2
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
milliseconds |  | 56.58 (54.478) | 87.22 (45.643)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -30.33, 95% CI 2-sided [-39.29 to -21.37] — Placebo minus Concerta

9. Secondary Outcome: Hour 5.5 Wide Range Assessment of Memory and Learning (WRAML-2) Finger Windows Backwards
Description: WRAML-2 (range: 0, 28) is designed to evaluate a child's ability to learn and to memorize information, consists of 9 subtests from which 4 summary indexes can be calculated: verbal memory index, visual memory index, learning index, and general memory index. During this test the investigator pointed to a longer and longer series of windows on a card at the rate of 1 location per second, and then the child was asked to reproduce the sequence exactly in reverse order. One point was given for each correctly recalled sequence, and the test was discontinued after 3 consecutive errors.
Time Frame: Hour 5.5 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Correct Sequences
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Correct Sequences |  | 9.8 (4.95) | 10.9 (4.5)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.0297, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -1.13, 95% CI 2-sided [-2.15 to -0.12] — Placebo minus Concerta

10. Secondary Outcome: Hour 5.5 Wide Range Assessment of Memory and Learning (WRAML-2) Finger Windows Forwards
Description: WRAML-2 (range: 0, 28) is designed to evaluate a child's ability to learn and to memorize information, consists of 9 subtests from which 4 summary indexes can be calculated: verbal memory index, visual memory index, learning index, and general memory index. During this test the investigator pointed to a longer and longer series of windows on a card at the rate of 1 location per second, and then the child was asked to reproduce the sequence exactly. One point was given for each correctly recalled sequence, and the test was discontinued after 3 consecutive errors.
Time Frame: Hour 5.5 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Correct Sequences
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Correct Sequences |  | 12.3 (4.94) | 13.2 (4.85)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.0955, Mixed Models Analysis — P-values were determined by using a general linear mixed model. Finger Windows Forwards was the first non-significant p-value in the gatekeeper sequence; Testing of additional endpoints in the sequence was still performed without any unqualified statements about the individual statistical significance; LS Mean Difference = -0.84, 95% CI 2-sided [-1.84 to 0.15] — Placebo minus Concerta

11. Secondary Outcome: Hour 5.5 Test of Variables of Attention (TOVA) Commissions
Description: The TOVA is a computerized, visual continuous performance test which provides measures of attention. The stimulus, presented for 100 milliseconds (ms) at the rate of 30 per minute, is a computer-presented square containing a square hole near the top (target) or bottom (non-target) edge. The first half of the TOVA requires that the child sustain attention while the second half requires inhibition of response to a non-target. Responses to non-targets. Higher score is preferable (observed range: -82.4, 128.9).
Time Frame: Hour 5.5 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Responses to non-targets
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Responses to non-targets |  | 78.35 (47.390) | 90.54 (36.132)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -14.37, 95% CI 2-sided [-21.52 to -7.23] — Placebo minus Concerta

12. Secondary Outcome: Hour 5.5 Wechsler Intelligence Scale for Children - 3rd ed. (WISC-III-PI) Digit Span Backwards
Description: Each child individually was given a sequence of numbers with the sequence becoming progressively longer. The child was then asked to repeat the digits in the same sequence, either forwards or backwards. Each sequence length was attempted twice. The test was complete after failure on both trials of any sequence length. One point was awarded if the participant passed only 1 trial of a sequence length. Zero points were given if the participant failed both trials. The maximum raw scores were 16 forwards and 14 backwards. A higher score was indicative of better recall and attention (range: 0, 14).
Time Frame: Hour 5.5 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Correct Sequences
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Correct Sequences |  | 4.8 (1.85) | 5.1 (1.87)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.2335, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -0.26, 95% CI 2-sided [-0.70 to 0.17] — Placebo minus Concerta

13. Secondary Outcome: Hour 8.75 Gray Silent Reading Test (GSRT)
Description: Gray Silent Reading Test (GSRT) is a reliable, validated measure of reading comprehension administered in the group setting during the first half hour of the homework session (observed range: 0, 141). A higher score is preferable as it means more questions were answered correctly.
Time Frame: Hour 8.75 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 89.1 (19.44) | 92.1 (19.03)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.2321, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -2.51, 95% CI 2-sided [-6.67 to 1.65] — Placebo minus Concerta

14. Secondary Outcome: Hour 7.5 Test of Handwriting Skills (Revised) (THS-R)
Description: The THS-R is a standardized, untimed assessment designed to evaluate neurosensory integration manifested in manuscript and cursive writing. The test includes the 10 subtests: writing from memory the upper- and lower-case letters of the alphabet in order, writing from dictation the upper and lower-case letters of the alphabet out of order, single digit-numbers out of order, selected words, and copying selected letters, words, and sentences. Each subtest was scored from zero (poorly formed letters) to 3 (perfectly formed letters). A higher score was preferable (observed range: 0, 118).
Time Frame: Hour 7.5 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 79.1 (13.86) | 82.7 (13.34)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -3.52, 95% CI 2-sided [-5.64 to -1.40] — Placebo minus Concerta

15. Secondary Outcome: Hour 3.5 Dynamic Indicators of Basic Early Literacy Skills (DIBELS)
Description: The DIBELS (observed range: 0, 212), used to assess reading fluency, consists of standardized, individually administered measures of early literacy development. These short (1 minute) fluency measures were developed based upon essential early literacy domains to assess development of phonological awareness, alphabetic understanding, and automaticity and fluency. Only the paragraph fluency component of an age/grade-appropriate DIBELS was used. Children read 3 stories and completed the forms. A higher score was preferable and indicated a greater number of words read correctly in the time allowed
Time Frame: Hour 3.5 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 110.8 (39.21) | 117.8 (39.38)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.0101, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -5.38, 95% CI 2-sided [-9.43 to -1.33] — Placebo minus Concerta

16. Secondary Outcome: Hour 5.5 Wechsler Intelligence Scale for Children - 3rd ed. (WISC-III-PI) Digit Span Forwards
Description: Each child individually was given a sequence of numbers with the sequence becoming progressively longer. The child was then asked to repeat the digits in the same sequence, either forwards or backwards. Each sequence length was attempted twice. The test was complete after failure on both trials of any sequence length. One point was awarded if the participant passed only 1 trial of a sequence length. Zero points were given if the participant failed both trials. The maximum raw scores were 16 forwards and 14 backwards. A higher score was indicative of better recall and attention (range: 0, 16).
Time Frame: Hour 5.5 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Correct Sequences
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Correct Sequences |  | 8.4 (1.60) | 8.5 (1.56)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.6642, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -0.09, 95% CI 2-sided [-0.53 to 0.34] — Placebo minus Concerta

17. Secondary Outcome: Hour 5.5 Test of Variables of Attention (TOVA) Omissions
Description: The TOVA is a computerized, visual continuous performance test which provides measures of attention. The stimulus, presented for 100 milliseconds (ms) at the rate of 30 per minute, is a computer-presented square containing a square hole near the top (target) or bottom (non-target) edge. The first half of the TOVA requires that the child sustain attention while the second half requires inhibition of response to a non-target. Number of targets missed. Higher score is preferable (observed range: -419.4, 108.9).
Time Frame: Hour 5.5 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Targets missed
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Targets missed |  | 36.34 (103.888) | 71.49 (82.508)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.0040, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -35.30, 95% CI 2-sided [-58.89 to -11.71] — Placebo minus Concerta

18. Secondary Outcome: Hour 3.0 Grammar Task
Description: This task, presented once during a laboratory school day, was designed to index "attention to detail" by determining how many grammatical mistakes each child could identify and circle in a brief paragraph. The errors were not difficult to identify and were designed to show attention to task, not comprehension. A higher number of errors identified, of those possible, was indicative of better attention - identification of grammatical errors (range: 0, 1 represents correct responses divided by the number of possible responses).
Time Frame: Hour 3.0 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 0.252 (0.1894) | 0.340 (0.2195)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -0.08, 95% CI 2-sided [-0.14 to -0.03] — Placebo minus Concerta

19. Secondary Outcome: Hour 8.75 Packet Activity - Short Story With Questions for Comprehension
Description: Packet Activities: Assessment of ability to organize, listen to instructions, initiate task, complete task, and distractibility, by completing a word search, reading a short story for comprehension on a multiple choice test, reading a longer story for comprehension on a true/false test, decoding a mystery sentence, and completing various vocabulary assessments (word choice, homophones; base/root words, alphabetic order)(range: 0, 1 represents correct responses divided by the number of possible responses).
Time Frame: Hour 8.75 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 0.619 (0.2435) | 0.699 (0.2239)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.0051, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -0.07, 95% CI 2-sided [-0.12 to -0.02] — Placebo minus Concerta

20. Secondary Outcome: Hour 8.75 Packet Activity - Identiy Root Word
Description: Packet Activities: Assessment of ability to organize, listen to instructions, initiate task, complete task, and distractibility, by completing a word search, reading a short story for comprehension on a multiple choice test, reading a longer story for comprehension on a true/false test, decoding a mystery sentence, and completing various vocabulary assessments (word choice, homophones; base/root words, alphabetic order) (range: 0, 1 represents correct responses divided by the number of possible responses).
Time Frame: Hour 8.75 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 0.580 (0.3478) | 0.638 (0.3230)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.1768, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -0.05, 95% CI 2-sided [-0.13 to 0.02] — Placebo minus Concerta

21. Secondary Outcome: Hour 8.75 Packet Activity - Alphabetize List of Words
Description: as for outcome 20
Time Frame: Hour 8.75 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 0.638 (0.3269) | 0.660 (0.3396)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.4245, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -0.02, 95% CI 2-sided [-0.09 to 0.04] — Placebo minus Concerta

22. Secondary Outcome: Hour 8.75 Packet Activity - Identify Multiple Meanings for Words
Description: as for outcome 20
Time Frame: Hour 8.75 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 0.814 (0.2936) | 0.821 (0.2839)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.9729, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean DIfference = 0.00, 95% CI 2-sided [-0.09 to 0.09] — Placebo minus Concerta

23. Secondary Outcome: Hour 8.75 Packet Activity - Complete Sentences Using Words Provided
Description: as for outcome 20
Time Frame: Hour 8.75 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 0.730 (0.3101) | 0.781 (0.2926)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.3486, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -0.04, 95% CI 2-sided [-0.12 to 0.04] — Placebo minus Concerta

24. Secondary Outcome: Hour 8.75 Packet Activity - Word Search
Description: as for outcome 20
Time Frame: Hour 8.75 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 0.955 (0.1272) | 0.984 (0.0862)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.1466, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = -0.03, 95% CI 2-sided [-0.07 to 0.01] — Placebo minus Concerta

25. Secondary Outcome: Hour 8.75 Packet Activity - Decode the Mystery Sentence
Description: as for outcome 20
Time Frame: Hour 8.75 of the Lab School Day During the Double-Blind Assessment Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Concerta: Chilfdren randomized to receive Concerta at lab school day 1 or lab school day 2
Arm/Group | Not Randomized | Placebo | Concerta
Number analyzed (Participants) | 0 | 64 | 67
Units on a scale |  | 0.989 (0.0278) | 0.955 (0.1661)
Statistical Analysis 1: Comparison: Placebo vs Concerta; Test type: Superiority or Other; p = 0.1368, Mixed Models Analysis — P-values were determined by using a general linear mixed model; LS Mean Difference = 0.03, 95% CI 2-sided [-0.01 to 0.08] — Placebo minus Concerta

ADVERSE EVENTS:
Time Frame: The sponsor collects adverse events for 14 weeks starting with the signing of the informed consent (up to 4 weeks prior to treatment) continuing until the final visit at early discontinuation or study completion (up to 10 weeks after start of treatment).
Groups:
- Placebo: Placebo was received during the lab school day
- Concerta: Concerta was received during the lab school day
- Open Label: dose adjustment period and double blind period other than lab school day
Arm/Group | Placebo | Concerta | Open Label
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67 | 0/89
Other Adverse Events (participants affected / at risk) | 5/67 | 9/67 | 75/89
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=67) | Concerta (N=67) | Open Label (N=89)
Initial insomnia (Psychiatric disorders) | 0 | 0 | 26
Affect lability (Psychiatric disorders) | 0 | 0 | 14
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 25
Vomiting (Gastrointestinal disorders) | 0 | 0 | 7
Nausea (Gastrointestinal disorders) | 0 | 0 | 6
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 20
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 12
Headache (Nervous system disorders) | 2 | 4 | 29
Irritability (General disorders) | 0 | 0 | 11
Fatigue (General disorders) | 0 | 0 | 7
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 9
Pharyngitis (Infections and infestations) | 0 | 0 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 9
Weight decreased (Investigations) | 0 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No